CLINICAL TRIAL: NCT01626872
Title: Long-Term Extension Study of MP-214 in Patients With Schizophrenia
Brief Title: Long-Term Study of MP-214 in Patients With Schizophrenia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A002-A5
Record Dates: First submitted 2012-06-19; First posted 2012-06-25 (Estimated); Results first posted 2021-04-12 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Antipsychotic Agents; Mental Disorder; Psychotropic Drugs; Dopamine Agents; Risperidone; Central Nervous System Agents
MeSH Terms: conditions — Schizophrenia; Mental Disorders | interventions — Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- MP-214 3mg (Experimental)
  Interventions: Drug: MP-214 3mg
- MP-214 6mg (Experimental)
  Interventions: Drug: MP-214 6mg
- MP-214 9mg (Experimental)
  Interventions: Drug: MP-214 9mg
- Risperidone 4mg (Active Comparator)
  Interventions: Drug: Risperidone 4mg

INTERVENTIONS:
Drug: MP-214 3mg — In the double-blind period (before Week 6), participants continue in the same arm they were on in core trial A002-A4 (except placebo arm starts 3mg or 6mg of MP-214). In the open-label period (after Week 6), patients will be rerandomized to 3mg or 6mg of MP-214. After the fourth week of the open-label treatment period, they will be received MP-214 at flexible doses (3mg or 6mg or 9mg).
  Arms: MP-214 3mg
Drug: MP-214 6mg — In the double-blind period (before Week 6), participants continue in the same arm they were on in core trial A002-A4 (except placebo arm starts 3mg or 6mg of MP-214). In the open-label period (after Week 6), patients will be rerandomized to 3mg or 6mg of MP-214. After the fourth week of the open-label treatment period, they will be received MP-214 at flexible doses (3mg or 6mg or 9mg).
  Arms: MP-214 6mg
Drug: MP-214 9mg — In the double-blind period (before Week 6), participants continue in the same arm they were on in core trial A002-A4 (except placebo arm starts 3mg or 6mg of MP-214). In the open-label period (after Week 6), patients will be rerandomized to 3mg or 6mg of MP-214. After the fourth week of the open-label treatment period, they will be received MP-214 at flexible doses (3mg or 6mg or 9mg).
  Arms: MP-214 9mg
Drug: Risperidone 4mg — In the double-blind period (before Week 6), participants continue in the same arm they were on in core trial A002-A4. In the open-label period (after Week 6), patients will be rerandomized to 3mg or 6mg of MP-214. After the fourth week of the open-label treatment period, they will be received MP-214 at flexible doses (3mg or 6mg or 9mg).
  Arms: Risperidone 4mg

SUMMARY:
The objective of this study is to evaluate the long-term safety, tolerability, and efficacy of MP-214 in patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the patient before the completion of Study A002-A4
* Patients who have completed the A002-A4 study

Exclusion Criteria:

* Patients who are experiencing ongoing, uncontrolled, clinically significant adverse events (AEs), as judged by the investigator (or subinvestigator)

The information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2012-09; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Sapporo, Hokkaido, Japan
- Seoul, South Korea
- Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Six patients who did not receive MP-214 during the open-label phase were excluded from the analysis population.
Period: Overall Study
Arm/Group | MP-214 3mg | MP-214 6mg | MP-214 9mg
Started | 81 | 109 | 58
Completed | 29 | 43 | 34
Not Completed | 52 | 66 | 24
Not completed — Physician Decision | 13 | 9 | 6
Not completed — Withdrawal by Subject | 19 | 27 | 8
Not completed — Adverse Event (including Death) | 20 | 28 | 8
Not completed — Protocol Violation (including Pregnancy) | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MP-214 3mg | MP-214 6mg | MP-214 9mg | Total
Number analyzed (Participants) | 81 | 109 | 58 | 248
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.0 (11.1) | 40.8 (11.3) | 42.5 (8.9) | 40.3 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 56 | 20 | 116
  Male | 41 | 53 | 38 | 132

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: The Numbers show Subjects with at least one Adverse Event
Time Frame: Up to 60 weeks (Treatment Period (48 weeks) and Follow-up Period (12 weeks))
Measure: Count of Participants; unit: Participants
Arm/Group | MP-214 3mg | MP-214 6mg | MP-214 9mg
Number analyzed (Participants) | 81 | 109 | 58
Participants | 67 | 92 | 50

ADVERSE EVENTS:
Arm/Group | MP-214 3mg | MP-214 6mg | MP-214 9mg
Serious Adverse Events (participants affected / at risk) | 14/81 | 33/109 | 14/58
Other Adverse Events (participants affected / at risk) | 55/81 | 72/109 | 42/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MP-214 3mg (N=81) | MP-214 6mg (N=109) | MP-214 9mg (N=58)
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1 | 0
Scar (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin scar contracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 2
Mania (Psychiatric disorders) | 1 | 0 | 0
Psychiatric symptom (Psychiatric disorders) | 0 | 1 | 0
Schizophrenia (Psychiatric disorders) | 9 | 26 | 11
Schizophrenia, paranoid type (Psychiatric disorders) | 1 | 1 | 1
Somatoform disorder (Psychiatric disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 2 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Abortion induced (Surgical and medical procedures) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MP-214 3mg (N=81) | MP-214 6mg (N=109) | MP-214 9mg (N=58)
Abdominal discomfort (Gastrointestinal disorders) | 1 | 3 | 3
Constipation (Gastrointestinal disorders) | 9 | 5 | 6
Dental caries (Gastrointestinal disorders) | 3 | 1 | 4
Diarrhoea (Gastrointestinal disorders) | 3 | 4 | 5
Nausea (Gastrointestinal disorders) | 4 | 2 | 4
Vomiting (Gastrointestinal disorders) | 5 | 3 | 4
Nasopharyngitis (Infections and infestations) | 21 | 13 | 13
Tinea pedis (Infections and infestations) | 0 | 3 | 6
Contusion (Injury, poisoning and procedural complications) | 3 | 5 | 3
Excoriation (Injury, poisoning and procedural complications) | 1 | 1 | 3
Blood creatine phosphokinase increased (Investigations) | 1 | 7 | 0
Weight increased (Investigations) | 4 | 11 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 4
Akathisia (Nervous system disorders) | 15 | 15 | 2
Dizziness (Nervous system disorders) | 4 | 6 | 2
Extrapyramidal disorder (Nervous system disorders) | 8 | 7 | 4
Headache (Nervous system disorders) | 9 | 7 | 4
Somnolence (Nervous system disorders) | 2 | 6 | 1
Tremor (Nervous system disorders) | 0 | 5 | 4
Anxiety (Psychiatric disorders) | 3 | 7 | 2
Insomnia (Psychiatric disorders) | 4 | 12 | 8
Restlessness (Psychiatric disorders) | 1 | 4 | 3
Schizophrenia (Psychiatric disorders) | 12 | 12 | 11
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3
Eczema (Skin and subcutaneous tissue disorders) | 1 | 5 | 6
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Hypertension (Vascular disorders) | 3 | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other